CLINICAL TRIAL: NCT00645879
Title: Safety & Efficacy of Investigational Products: Ornithine Alpha-ketoglutarate, Glutamine, or Disodium Citrate on Hyperammonemia in Propionic Acidemia.
Brief Title: Anaplerotic Therapy in Propionic Acidemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Nicola Longo (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor-Investigator, Nicola Longo, MD, Professor, Biochemical Geneticist, University of Utah
Organization: University of Utah (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 24806; 1R21DK077415-01A1 (NIH); ANA-PA-001 (Other: University of Utah)
Record Dates: First submitted 2008-03-25; First posted 2008-03-28 (Estimated); Last update posted 2015-01-21 (Estimated); Status verified 2015-01

CONDITIONS: Propionic Acidemia
Keywords: Propionic Acidemia; hyperammonemia; hypotonia; glutamine; ornithine alpha ketoglutarate; citrate
MeSH Terms: conditions — Propionic Acidemia; Hyperammonemia; Muscle Hypotonia | interventions — ornithine alpha-ketoglutarate; Glutamine; Glutamic Acid; Sodium Citrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- OKG, Glutamine, and Disodium Citrate (Experimental): Ornithine Alpha Ketoglutarate for 4 weeks, followed by 2 week washout period. 4 weeks Glutamine, followed by 2 week washout period. 4 weeks Disodium Citrate, followed by 2 to 12 week washout period. Then continue an additional 30 weeks on Disodium Citrate (drug producing the best increment in plasma glutamine levels).
  Interventions: Drug: ornithine alpha ketoglutarate; Drug: glutamine; Drug: disodium citrate

INTERVENTIONS:
Drug: ornithine alpha ketoglutarate — A dose of 400 mg/kg up to 16 g per day was selected. Split into 2 doses taken for 4 weeks. If determined the drug with the best effect, drug will be taken for 30 weeks.
  Other Names: OKG
Drug: glutamine — A dose of 400 mg/kg up to 16 g per day was selected. Split into 2 doses taken for 4 weeks. If determined the drug with the best effects, drug will be taken for 30 weeks.
  Other Names: Glutamic Acid
Drug: disodium citrate — Dose: 7.5 mEq/Kg or 658 mg/kg up to 16 g per day Split into 2 doses taken for 4 weeks. If determined the drug with the best effects, drug will be taken for 30 weeks.
  Other Names: Citric Acid Sodium Salt, Sodium Citrate

SUMMARY:
The objective of this project is to define whether nutritional supplements (ornithine alpha-ketoglutarate, glutamine, or citrate) capable of filling-up the citric acid cycle (anaplerotic therapy) can improve hyperammonemia, glutamine levels, and outcome in patients with propionic acidemia. Ornithine alpha-ketoglutarate, glutamine, and citrate are commonly used as nutritional supplements specially by athletes to increase muscle strength. They can be mixed with formula or other foods.

DETAILED DESCRIPTION:
Propionic acidemia is caused by deficiency of propionyl CoA carboxylase that impairs the supply of succinyl CoA to the citric acid (Krebs) cycle. The Krebs cycle is responsible for obtaining energy from food in the form of ATP. ATP is essential for muscle contraction and correct functioning of all organs including the hearth, the kidney, and the pancreas.

Patients with propionic acidemia develop hyperammonemia at birth that recurs during episodes of metabolic decompensation. We found that plasma levels of the amino acids glutamine/glutamate are reduced in patients with propionic acidemia and decrease, rather than increase (like in urea cycle defects or other types of hyperammonemia) with hyperammonemia. Since alpha-ketoglutarate is the main source of endogenous glutamate/glutamine synthesis, our hypothesis is that chronic hyperammonemia and progressive dysfunction of multiple organs in patients with propionic acidemia is due to a functional insufficiency of the citric acid (Krebs) cycle with defective production of alpha-ketoglutarate. The basic deficiency of intermediates of the Krebs cycle can decrease production of ATP and explain the low muscle tone, progressive organ dysfunction, and poor long-term outcome of patients with propionic acidemia.

To test this hypothesis, we will test whether dietary supplementation with alpha ketoglutarate precursors (in the form of ornithine alpha ketoglutarate, glutamine or citrate) can improve plasma ammonia and overall outcome in patients with propionic acidemia. In this study, a limited number of patients (3) with propionic acidemia will be given the 3 different nutritional supplements and studied at regular intervals to see whether their glutamine/glutamate levels improve and if they have fewer episodes of hyperammonemia or acute decompensation. The supplement that produces the best increase in plasma glutamine levels will be tested for an additional 30 weeks. Children's development and motor skills will be tested before and after therapy to see if there is any improvement. The study will be conducted on outpatients at the University of Utah Clinical Research Center. If the initial trial is successful, we will try to launch a national trial involving multiple centers in the US and abroad to involve the largest number of patients possible.

The current therapy of propionic acidemia is based on restriction of precursors of propionic acid (methionine, valine, isoleucine, threonine, odd chain fatty acids, cholesterol) and administration of carnitine to help remove toxic organic acids. This therapy is not effective in preventing the long-term complications of the disease, even in children identified at birth by newborn screening. This research will test a completely new way of treating patients with severe and disabling metabolic disorders using replacement of downstream products involved in the generation of energy (ATP). This approach, if effective, could be extended to a number of other diseases, including other organic acidemias and mitochondrial disorders.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of propionic acidemia (propionyl CoA carboxylase deficiency)

Exclusion Criteria:

* Severe illness with cardiac or hepatic compromise that could affect study results
* Use of other investigative therapies
* Inability to comply with study directions

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 3 (Actual)
Dates: Start 2008-07; Primary Completion 2009-08 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Define safety and efficacy of nutritional therapy with these investigational products: L-Ornithine alpha-ketoglutarate, Glutamine, or disodium citrate (anaplerotic therapy) on hyperammonemia and outcome in patients with propionic acidemia. | end of study

SECONDARY OUTCOMES:
Define the effect of citrate, alpha-ketoglutarate and glutamine on plasma amino acids, acylcarnitines, ammonia, lactic acid and urine organic acids in patients with propionic acidemia. | end of study
Evaluate the effect of investigational products on the developmental quotient and medical complications in patients with propionic acidemia. | end of study

CONTACTS AND LOCATIONS:
Overall Officials: Nicola Longo, MD, PhD, Principal Investigator — University of Utah
Locations (1):
- University of Utah, Department of Pediatrics, Salt Lake City, Utah, United States

REFERENCES:
- [Background] Deodato F, Boenzi S, Santorelli FM, Dionisi-Vici C. Methylmalonic and propionic aciduria. Am J Med Genet C Semin Med Genet. 2006 May 15;142C(2):104-12. doi: 10.1002/ajmg.c.30090. PMID 16602092
- [Background] Dionisi-Vici C, Deodato F, Roschinger W, Rhead W, Wilcken B. 'Classical' organic acidurias, propionic aciduria, methylmalonic aciduria and isovaleric aciduria: long-term outcome and effects of expanded newborn screening using tandem mass spectrometry. J Inherit Metab Dis. 2006 Apr-Jun;29(2-3):383-9. doi: 10.1007/s10545-006-0278-z. PMID 16763906
- [Background] Mochel F, DeLonlay P, Touati G, Brunengraber H, Kinman RP, Rabier D, Roe CR, Saudubray JM. Pyruvate carboxylase deficiency: clinical and biochemical response to anaplerotic diet therapy. Mol Genet Metab. 2005 Apr;84(4):305-12. doi: 10.1016/j.ymgme.2004.09.007. PMID 15781190
- [Background] Roe CR, Sweetman L, Roe DS, David F, Brunengraber H. Treatment of cardiomyopathy and rhabdomyolysis in long-chain fat oxidation disorders using an anaplerotic odd-chain triglyceride. J Clin Invest. 2002 Jul;110(2):259-69. doi: 10.1172/JCI15311. PMID 12122118
- [Background] Filipowicz HR, Ernst SL, Ashurst CL, Pasquali M, Longo N. Metabolic changes associated with hyperammonemia in patients with propionic acidemia. Mol Genet Metab. 2006 Jun;88(2):123-30. doi: 10.1016/j.ymgme.2005.11.016. Epub 2006 Jan 10. PMID 16406646
- [Derived] Longo N, Price LB, Gappmaier E, Cantor NL, Ernst SL, Bailey C, Pasquali M. Anaplerotic therapy in propionic acidemia. Mol Genet Metab. 2017 Sep;122(1-2):51-59. doi: 10.1016/j.ymgme.2017.07.003. Epub 2017 Jul 12. PMID 28712602